CLINICAL TRIAL: NCT05477030
Title: Effect of Automated Insulin Delivery With Advanced Closed-loop on Glucose Outcomes and Early-stage Diabetic Complications
Brief Title: Effect of Automated Insulin Delivery on Early-stage Diabetic Complications
Acronym: AID-Comp
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Paolo Fiorina, MD, MD, Ph.D, Full Professor, University of Milan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022004
Record Dates: First submitted 2022-06-16; First posted 2022-07-28 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Type 1 Diabetes
Keywords: Automated insulin delivery; Type 1 Diabetes complications
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Open label randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Group A (Intervention) (Active Comparator): Group treated with automated insulin delivery (advanced hybrid closed-loop)
  Interventions: Device: Medtronic MiniMed 780G with SmartGuard activation
- Study Group B (Control) (Active Comparator): Group treated with predictive low glucose suspend (sensor augmented pump - PLGS)
  Interventions: Device: Medtronic MiniMed 780G without SmartGuard activation

INTERVENTIONS:
Device: Medtronic MiniMed 780G with SmartGuard activation — Insulin pump implemented with alghoritm for automatic modulation of insulin delivery (to increase time in glucose range 70-180 mg/dl)
  Arms: Study Group A (Intervention)
Device: Medtronic MiniMed 780G without SmartGuard activation — Insulin pump implemented with alghoritm for low glucose insulin suspension (to reduce hypoglycemia rate)
  Arms: Study Group B (Control)

SUMMARY:
Aim of this study is to verify the effects of an advanced HCL (Medtronic Minimed™ 780G) compared to SAP with PLGS on metabolic outcomes and markers of early microvascular damage in a population of adults with T1D previously treated with CSII. Evaluation of endothelial disfunction and autonomic neuropathy will also be performed.

DETAILED DESCRIPTION:
New algorithms for the automation of insulin delivery (AID) are showing great benefit on glucose control in people with type 1 diabetes. Indeed, Hybrid closed loop (HCL) systems can improve HbA1c levels, percentage of time in defined glucose range, time below range and time over range, according to RCT and observational studies results. However, scientific evidences demonstrating potential benefits on the reduction of diabetes complications are limited regarding CSII or SAP with demonstrated reduction of cardiovascular mortality, improvement of albuminuria and peripheral nerve damage.

Data on AID effects on complications of diabetes are missing. In this study intermediate damage markers will be measured to assess potential effects of AID in comparison to sensor augmented pumps.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients
* T1D patients above 18 years in CSII treatment for at least 3 months
* HbA1c values between 6.0% and 9.5%
* Disease duration ≥ 2 years
* Written informed consent obtained from the patient

Exclusion Criteria:

* Pregnancy
* Participation to other clinical trials
* A history of alcohol or drug abuse
* Advanced diabetic nephropathy defined as presence of albuminuria ≥ 300 mg/g or eGFR < 60 ml/min/1,73m2
* Proliferative Diabetic retinopathy or macular edema
* Established Atherosclerotic Cardiovascular Disease (ASCVD) or history of heart failure
* Presence of serious diseases or conditions which in the opinion of the Investigator makes patient non-eligible for the study
* Hypoglycemia Unawareness (Clarke score > 4)
* Patients unable to understand spoken and written Italian language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2022-02-23 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2024-02-23 (Estimated)

PRIMARY OUTCOMES:
Time in glycemic range 70-180 mg/dl | From Baseline to 26 weeks
  time spent by the patient in glucose range
Glycated Hemoglobin (HbA1c) | From Baseline to 26 weeks
  percentage of hemoglobin glycosylated

SECONDARY OUTCOMES:
Early microangiopathic damage markers: sTNFR-1/2 | From Baseline to 26 weeks
  sTNFR-1/2 (pg/ml)
Early microangiopathic damage markers: B-2 microglobulin | From Baseline to 26 weeks
  B-2 microglobulin (pg/ml)
Early microangiopathic damage markers: cystatin C | From Baseline to 26 weeks
  cystatin C (ng/ml)
Early microangiopathic damage markers: neutrophil gelatinase-associated lipocalin | From Baseline to 26 weeks
  neutrophil gelatinase-associated lipocalin (ng/ml)
Early microangiopathic damage markers: osteopontin | From Baseline to 26 weeks
  osteopontin (pg/ml)
Early microangiopathic damage markers: vWF levels | From Baseline to 26 weeks
  vWF levels (ng/ml)
Endothelial disfunction | From Baseline to 26 weeks
  Endothelial-dependent dilation (EDD) is considered a marker of dysfunctional abnormalities involved in early phases of atherosclerosis development. Changes in EDD precede structural changes and occurs in the preclinical phase of vascular disease.
  In the present study endothelial dependent dilation is assessed by color Doppler evaluation of flow increase after hyperemia.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Fiorina, MD, PhD, Principal Investigator — ASST-FBF-Sacco, University of Milan
Locations (1):
- ASST FBF Sacco, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Diabetes Control and Complications Trial Research Group; Nathan DM, Genuth S, Lachin J, Cleary P, Crofford O, Davis M, Rand L, Siebert C. The effect of intensive treatment of diabetes on the development and progression of long-term complications in insulin-dependent diabetes mellitus. N Engl J Med. 1993 Sep 30;329(14):977-86. doi: 10.1056/NEJM199309303291401. PMID 8366922
- [Result] Writing Team for the Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications Research Group. Effect of intensive therapy on the microvascular complications of type 1 diabetes mellitus. JAMA. 2002 May 15;287(19):2563-9. doi: 10.1001/jama.287.19.2563. PMID 12020338
- [Result] Nathan DM, Cleary PA, Backlund JY, Genuth SM, Lachin JM, Orchard TJ, Raskin P, Zinman B; Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications (DCCT/EDIC) Study Research Group. Intensive diabetes treatment and cardiovascular disease in patients with type 1 diabetes. N Engl J Med. 2005 Dec 22;353(25):2643-53. doi: 10.1056/NEJMoa052187. PMID 16371630
- [Result] Pettus JH, Zhou FL, Shepherd L, Preblick R, Hunt PR, Paranjape S, Miller KM, Edelman SV. Incidences of Severe Hypoglycemia and Diabetic Ketoacidosis and Prevalence of Microvascular Complications Stratified by Age and Glycemic Control in U.S. Adult Patients With Type 1 Diabetes: A Real-World Study. Diabetes Care. 2019 Dec;42(12):2220-2227. doi: 10.2337/dc19-0830. Epub 2019 Sep 23. PMID 31548241
- [Result] Pickup JC, Sutton AJ. Severe hypoglycaemia and glycaemic control in Type 1 diabetes: meta-analysis of multiple daily insulin injections compared with continuous subcutaneous insulin infusion. Diabet Med. 2008 Jul;25(7):765-74. doi: 10.1111/j.1464-5491.2008.02486.x. PMID 18644063
- [Result] Pankowska E, Blazik M, Dziechciarz P, Szypowska A, Szajewska H. Continuous subcutaneous insulin infusion vs. multiple daily injections in children with type 1 diabetes: a systematic review and meta-analysis of randomized control trials. Pediatr Diabetes. 2009 Feb;10(1):52-8. doi: 10.1111/j.1399-5448.2008.00440.x. Epub 2008 Aug 27. PMID 18761648
- [Result] EQuality1 Study Group--Evaluation of QUALITY of Life and Costs in Diabetes Type 1; Nicolucci A, Maione A, Franciosi M, Amoretti R, Busetto E, Capani F, Bruttomesso D, Di Bartolo P, Girelli A, Leonetti F, Morviducci L, Ponzi P, Vitacolonna E. Quality of life and treatment satisfaction in adults with Type 1 diabetes: a comparison between continuous subcutaneous insulin infusion and multiple daily injections. Diabet Med. 2008 Feb;25(2):213-20. doi: 10.1111/j.1464-5491.2007.02346.x. Epub 2008 Jan 14. PMID 18201210
- [Result] Maniatis AK, Toig SR, Klingensmith GJ, Fay-Itzkowitz E, Chase HP. Life with continuous subcutaneous insulin infusion (CSII) therapy: child and parental perspectives and predictors of metabolic control. Pediatr Diabetes. 2001 Jun;2(2):51-7. doi: 10.1034/j.1399-5448.2001.002002051.x. PMID 15016198
- [Result] Bergenstal RM, Tamborlane WV, Ahmann A, Buse JB, Dailey G, Davis SN, Joyce C, Perkins BA, Welsh JB, Willi SM, Wood MA; STAR 3 Study Group. Sensor-augmented pump therapy for A1C reduction (STAR 3) study: results from the 6-month continuation phase. Diabetes Care. 2011 Nov;34(11):2403-5. doi: 10.2337/dc11-1248. Epub 2011 Sep 20. PMID 21933908
- [Result] Forlenza GP, Li Z, Buckingham BA, Pinsker JE, Cengiz E, Wadwa RP, Ekhlaspour L, Church MM, Weinzimer SA, Jost E, Marcal T, Andre C, Carria L, Swanson V, Lum JW, Kollman C, Woodall W, Beck RW. Predictive Low-Glucose Suspend Reduces Hypoglycemia in Adults, Adolescents, and Children With Type 1 Diabetes in an At-Home Randomized Crossover Study: Results of the PROLOG Trial. Diabetes Care. 2018 Oct;41(10):2155-2161. doi: 10.2337/dc18-0771. Epub 2018 Aug 8. PMID 30089663
- [Result] Bergenstal RM, Garg S, Weinzimer SA, Buckingham BA, Bode BW, Tamborlane WV, Kaufman FR. Safety of a Hybrid Closed-Loop Insulin Delivery System in Patients With Type 1 Diabetes. JAMA. 2016 Oct 4;316(13):1407-1408. doi: 10.1001/jama.2016.11708. No abstract available. PMID 27629148
- [Result] Nimri R, Muller I, Atlas E, Miller S, Fogel A, Bratina N, Kordonouri O, Battelino T, Danne T, Phillip M. MD-Logic overnight control for 6 weeks of home use in patients with type 1 diabetes: randomized crossover trial. Diabetes Care. 2014 Nov;37(11):3025-32. doi: 10.2337/dc14-0835. Epub 2014 Jul 30. PMID 25078901
- [Result] Garg SK, Weinzimer SA, Tamborlane WV, Buckingham BA, Bode BW, Bailey TS, Brazg RL, Ilany J, Slover RH, Anderson SM, Bergenstal RM, Grosman B, Roy A, Cordero TL, Shin J, Lee SW, Kaufman FR. Glucose Outcomes with the In-Home Use of a Hybrid Closed-Loop Insulin Delivery System in Adolescents and Adults with Type 1 Diabetes. Diabetes Technol Ther. 2017 Mar;19(3):155-163. doi: 10.1089/dia.2016.0421. Epub 2017 Jan 30. PMID 28134564
- [Result] Salehi P, Roberts AJ, Kim GJ. Efficacy and Safety of Real-Life Usage of MiniMed 670G Automode in Children with Type 1 Diabetes Less than 7 Years Old. Diabetes Technol Ther. 2019 Aug;21(8):448-451. doi: 10.1089/dia.2019.0123. Epub 2019 Jun 5. PMID 31166801
- [Result] Lepore G, Scaranna C, Corsi A, Dodesini AR, Trevisan R. Switching from Suspend-Before-Low Insulin Pump Technology to a Hybrid Closed-Loop System Improves Glucose Control and Reduces Glucose Variability: A Retrospective Observational Case-Control Study. Diabetes Technol Ther. 2020 Apr;22(4):321-325. doi: 10.1089/dia.2019.0302. Epub 2020 Feb 11. PMID 31617752
- [Result] Steineck I, Cederholm J, Eliasson B, Rawshani A, Eeg-Olofsson K, Svensson AM, Zethelius B, Avdic T, Landin-Olsson M, Jendle J, Gudbjornsdottir S; Swedish National Diabetes Register. Insulin pump therapy, multiple daily injections, and cardiovascular mortality in 18,168 people with type 1 diabetes: observational study. BMJ. 2015 Jun 22;350:h3234. doi: 10.1136/bmj.h3234. PMID 26100640
- [Result] Rosenlund S, Hansen TW, Rossing P, Andersen S. Effect of Sensor-Augmented Pump Treatment Versus Multiple Daily Injections on Albuminuria: A 1-Year Randomized Study. J Clin Endocrinol Metab. 2015 Nov;100(11):4181-8. doi: 10.1210/jc.2015-2839. Epub 2015 Sep 21. PMID 26390102
- [Result] Rosenlund S, Hansen TW, Andersen S, Rossing P. Effect of 4 years subcutaneous insulin infusion treatment on albuminuria, kidney function and HbA1c compared with multiple daily injections: a longitudinal follow-up study. Diabet Med. 2015 Nov;32(11):1445-52. doi: 10.1111/dme.12950. Epub 2015 Oct 6. PMID 26331364
- [Result] Zabeen B, Craig ME, Virk SA, Pryke A, Chan AK, Cho YH, Benitez-Aguirre PZ, Hing S, Donaghue KC. Insulin Pump Therapy Is Associated with Lower Rates of Retinopathy and Peripheral Nerve Abnormality. PLoS One. 2016 Apr 6;11(4):e0153033. doi: 10.1371/journal.pone.0153033. eCollection 2016. PMID 27050468
- [Result] Battelino T, Danne T, Bergenstal RM, Amiel SA, Beck R, Biester T, Bosi E, Buckingham BA, Cefalu WT, Close KL, Cobelli C, Dassau E, DeVries JH, Donaghue KC, Dovc K, Doyle FJ 3rd, Garg S, Grunberger G, Heller S, Heinemann L, Hirsch IB, Hovorka R, Jia W, Kordonouri O, Kovatchev B, Kowalski A, Laffel L, Levine B, Mayorov A, Mathieu C, Murphy HR, Nimri R, Norgaard K, Parkin CG, Renard E, Rodbard D, Saboo B, Schatz D, Stoner K, Urakami T, Weinzimer SA, Phillip M. Clinical Targets for Continuous Glucose Monitoring Data Interpretation: Recommendations From the International Consensus on Time in Range. Diabetes Care. 2019 Aug;42(8):1593-1603. doi: 10.2337/dci19-0028. Epub 2019 Jun 8. PMID 31177185
- [Result] Fiorina P, La Rocca E, Venturini M, Minicucci F, Fermo I, Paroni R, D'Angelo A, Sblendido M, Di Carlo V, Cristallo M, Del Maschio A, Pozza G, Secchi A. Effects of kidney-pancreas transplantation on atherosclerotic risk factors and endothelial function in patients with uremia and type 1 diabetes. Diabetes. 2001 Mar;50(3):496-501. doi: 10.2337/diabetes.50.3.496. PMID 11246868
- [Result] Zoppini G, Bergamini C, Trombetta M, Sabbagh L, Dauriz M, Mantovani A, Targher G, Fossa I, Rinaldi E, Bonora E. Increased aortic stiffness index in patients with type 1 diabetes without cardiovascular disease compared to controls. J Endocrinol Invest. 2019 Sep;42(9):1109-1115. doi: 10.1007/s40618-019-01032-7. Epub 2019 Mar 16. PMID 30877659
- [Result] Clarke WL, Cox DJ, Gonder-Frederick LA, Julian D, Schlundt D, Polonsky W. Reduced awareness of hypoglycemia in adults with IDDM. A prospective study of hypoglycemic frequency and associated symptoms. Diabetes Care. 1995 Apr;18(4):517-22. doi: 10.2337/diacare.18.4.517. PMID 7497862
- [Result] Polonsky WH, Fisher L, Earles J, Dudl RJ, Lees J, Mullan J, Jackson RA. Assessing psychosocial distress in diabetes: development of the diabetes distress scale. Diabetes Care. 2005 Mar;28(3):626-31. doi: 10.2337/diacare.28.3.626. PMID 15735199
- [Result] Bott U, Muhlhauser I, Overmann H, Berger M. Validation of a diabetes-specific quality-of-life scale for patients with type 1 diabetes. Diabetes Care. 1998 May;21(5):757-69. doi: 10.2337/diacare.21.5.757. PMID 9589237